CLINICAL TRIAL: NCT03536273
Title: The Effect of Pilates Group Exercise Program on Functional Movement Scores, Posture, Depression and Quality of Life in Sedentary Women
Brief Title: The Effect of Pilates Group Exercise Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Emre Serdar Vayvay, Lecturer, Medipol University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10840098-604.01.01-E.45484
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Sedentary Lifestyle
Keywords: sedentary; pilates exercises; functional movement screen; posture; quality of life
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Functional Movement Screen (Experimental)
  Interventions: Other: Pilates Group Exercises
- Posture Analysis (Experimental)
  Interventions: Other: Pilates Group Exercises
- Depression Level (Experimental)
  Interventions: Other: Pilates Group Exercises
- Quality of Life (Experimental)
  Interventions: Other: Pilates Group Exercises

INTERVENTIONS:
Other: Pilates Group Exercises — For 12 weeks, 3 repetitions per week

SUMMARY:
INTRODUCTION AND AIM: The Pilates exercises were introduced by Joseph Pilates in the 1920s, originally called 'centering'. These exercises work on 6 simple principles with or without special equipment. These principles are; centering, concentration, tenderness, flow and respiration. (Yamato et al., 2016) Functional movement analysis is a screening system developed by physiotherapist Gray Cook. Functional deficits of the person are detected by 7 different movements (Cook, Burton and Hoogenboom 2006a, Cook, Burton and Hoogenboom 2006b). In a single study they compared in the literature that assessed the effect of Pilates exercises on functional movement, this activity was explored on recreational runners (Laws, Williams and Wilson 2017). The aim of this study was to investigate the effect of 12-week pilates group exercise training on functional movement scores in sedentary women. Secondarily; posture, depression level and quality of life will be evaluated.

MATERIAL-METHODS: This study has been reviewed by Ethics Committee of Non-Interventional Researches of the University of Medipol in Istanbul and its ethical conformity has been approved. (10840098-604.01.01-E.45484). Participants were informed of the voluntary consent form and signed the consent form.

Participants 20 sedentary women were included in the study between 30-50 years of age.

Evaluations

Demographic information (Age, Occupation, Height, Weight) of the persons will be recorded.Functional Movement Analysis; Postural Analysis, Depression level; Health Related Life quality will be recorded.

Application Pilates exercises will be applied by a qualified physiotherapist with an internationally recognized certificate on the subject. Participants will be asked to come up with suitable outfits. the exercise room will be set at the ideal temperature and well ventilated. The exercises to be done in the form of group exercises will be started with an entry level, and the level of the exercises will be increased appropriately in the following weeks. Each group will consist of no more than 10 people and the exercises will continue for three sessions per week for 12 weeks. The evaluations will be repeated before exercise, at the end of 12 weeks of exercise and after 3 months from finish of the exercise period.

ELIGIBILITY:
Inclusion Criteria:

* Have not had a surgical operation involving the musculoskeletal system in the past six months.
* Not to have a systemic disease leading preventing from exercise.
* Not having had any exercise in the last 3 months.

Exclusion Criteria:

* Do not want to continue exercises.
* To feel pain, discomfort during tests.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Functional Movement Screen Total Score | 20 minutes
  7 subtests

SECONDARY OUTCOMES:
New York Posture Analysis Score | 10 min
  Observational scale filled by physiotherapist
Beck Depression Scale | 5 min
  Scale to be marked by the participant
Short Form 36 Quality of Life Assessment | 10 min
  Scale to be marked by the participant

CONTACTS AND LOCATIONS:
Overall Officials: Emre S Atalay, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Emre Serdar Atalay, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No